CLINICAL TRIAL: NCT05509270
Title: Assessing the Relative Efficacy of Communication Modalities for Messages Promoting Flu Shots
Brief Title: Efficacy of Communication Modalities for Promoting Flu Shots
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Christopher F Chabris, PhD, Professor, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0373
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Influenza Vaccination; Health Promotion; Health Behavior; Risk Reduction
Keywords: Flu Vaccine; Choice Architecture; Machine Learning; Perceived Credibility
MeSH Terms: conditions — Influenza, Human; Health Behavior; Risk Reduction Behavior | interventions — College Fraternities and Sororities; Patient Portals

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Providers who prescribe vaccination and diagnose conditions will not be randomized to study arms or informed of patient assignment. Although patients will not be explicitly informed which arm they have been randomized to, they will be aware of the messages they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (No Intervention): No additional pro-vaccination intervention - some patients are currently targeted for flu vaccination messages due to a non-machine learning-based assessment that they are at high risk for complications, but are not told that they are at high risk or that they have been targeted
- Letter only (Experimental): This group will receive a letter telling them they are at high risk for flu and complications
  Interventions: Behavioral: Letter
- Patient portal only (Experimental): This group will receive a patient portal message telling them they are at high risk for flu and complications
  Interventions: Behavioral: Patient portal
- SMS only (Experimental): This group will receive an SMS telling them they are at high risk for flu and complications
  Interventions: Behavioral: SMS
- Patient portal + SMS (Experimental): This group will receive a patient portal message and an SMS telling them they are at high risk for flu and complications
  Interventions: Behavioral: Patient portal; Behavioral: SMS
- Letter + Patient portal + SMS (Experimental): This group will receive a letter, a patient portal message, and an SMS telling them they are at high risk for flu and complications
  Interventions: Behavioral: Letter; Behavioral: Patient portal; Behavioral: SMS

INTERVENTIONS:
Behavioral: Letter — Mailed letter about flu vaccination
  Arms: Letter + Patient portal + SMS; Letter only
Behavioral: Patient portal — Patient portal message about flu vaccination
  Arms: Letter + Patient portal + SMS; Patient portal + SMS; Patient portal only
Behavioral: SMS — SMS about flu vaccination
  Arms: Letter + Patient portal + SMS; Patient portal + SMS; SMS only

SUMMARY:
The purpose of this study is to test which modalities (mailed letter, short message service [SMS] text, or patient portal messages) are most effective for encouraging flu shots in high-risk patients.

DETAILED DESCRIPTION:
The Centers for Disease Control (CDC) recommends a flu vaccination to everyone aged 6+ months, with rare exception; almost anyone can benefit from the vaccine, which can reduce illnesses, missed work, hospitalizations, and death. Flu shots are particularly important for patients at high risk of experiencing severe outcomes.

During the 2020-21 and 2021-22 flu seasons, the study team sent messages to Geisinger patients in the top 10% of risk for flu and complications according to an artificial intelligence algorithm. Messages that told patients they were at high risk significantly increased their likelihood of getting vaccinated.

The present study will extend previous work by testing which modality or modalities are most effective at boosting flu shot rates in patients at high risk. In previous campaigns, patients received messages via all communication modalities patients were eligible for (mailed letter, SMS text, and/or patient portal message). In this study, patients will be randomized to receive high-risk messages in one or more modalities.

ELIGIBILITY:
Inclusion Criteria:

* Included on a list of active Geisinger patients (all patients on this list attended at least one primary care appointment at Geisinger between 10/1/2008 and 4/13/2022, and either had a Geisinger primary care provider assigned as of April 2022, or were in the Electronic Health Record [EHR] since at least September 2021 and had at least one encounter in 2020-2022)
* Aged 18 or older
* In the top 10% of risk for flu and flu complications, according to Medial's flu complications machine learning algorithm (which operates on coded EHR data)
* Has a Geisinger PCP assigned as of August 2022
* Has had an encounter in the last 2 years as of August 2022

Exclusion Criteria:

- Cannot be contacted via any of the communication modalities (e.g., letter, patient portal, SMS) being used in the study, either due to insufficient/missing contact information in the EHR or because they opted out of all modalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43225 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Flu vaccination | 4 weeks after the first messages are sent in the study
  Flu vaccination within 4 weeks of the first message send date

OTHER OUTCOMES:
High confidence flu diagnosis | Up to 8 months
  Patient received a flu diagnosis via a positive polymerase chain reaction (PCR)/antigen/molecular test (yes/no) during the 2022-23 flu season (from the first message send date through April 30, 2023).
"Likely flu" diagnosis | Up to 8 months
  Received a "high confidence flu" diagnosis (with positive PCR/antigen/molecular test) and/or "likely flu" diagnosis (as assessed via International Classification of Disease [ICD] codes or Tamiflu administration or positive PCR/antigen/molecular test) (yes/no) during the 2022-23 flu season (from the first message send date through April 30, 2023).
  Note that "likely flu" is a superset of the "high confidence flu" diagnoses.
Flu complications | Up to 11 months
  Diagnosed with flu-related complications (yes/no) from the first message send date through July 31, 2023.
ER visits | Up to 11 months
  Number of ER visits from the first message send date through July 31, 2023.
Hospitalizations | Up to 11 months
  Number of hospitalizations from the first message send date through July 31, 2023.
COVID-19 vaccination rates | Up to 8 months
  Received at least one COVID-19 vaccination (yes/no) during the 2022-23 flu season (from the first message send date through April 30, 2023).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chabris, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT05509270/Prot_SAP_000.pdf